CLINICAL TRIAL: NCT00067795
Title: HIV Antigen-Specific Immune Responses - A Comparison of Alternative In Vitro Assays From Subjects Characterized as Either "Stable HAART" or "Efficient Immune Control"
Brief Title: Evaluating Immune Function Tests in People With HIV
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: ACTG A5181
Record Dates: First submitted 2003-08-27; First posted 2003-08-28 (Estimated); Last update posted 2010-11-22 (Estimated); Status verified 2010-11

CONDITIONS: HIV Infections
Keywords: Treatment Experienced; Antiretroviral Therapy, Highly Active; HIV Antigens; Cohort Studies; Immunity, Cellular; T-Lymphocytes
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Some people's immune systems are able to control HIV infection without anti-HIV drugs. Other people with HIV must take drugs to prevent the virus from destroying their immune systems. There are many different laboratory tests that measure immune function in people with HIV. This study will compare some of these tests to see if they consistently measure differences between people who control the HIV without anti-HIV drugs and those who must take drugs.

DETAILED DESCRIPTION:
The efficiency of the immune response to HIV antigens is the critical feature that allows some individuals with chronic HIV infection to maintain low level viremia (less than 3000 copies/ml). The fundamental measurement of this response is the steady state level of viremia in the absence of antiretroviral drugs. However, using this clinical endpoint in vaccine and drug trials is time-consuming. Several laboratory assays of HIV T cell function have been developed to measure the key characteristics of an efficient immune response. This study will evaluate these assays in two distinct patient populations.

Two patient cohorts will be followed in this study. Cohort A will enroll patients who are stable on highly active antiretroviral therapy (HAART). These patients will have been on the same HAART regimen for at least 9 months prior to study entry. Cohort B will enroll patients with chronic HIV infection and efficient immune control. These patients will have not been on any antiretroviral drugs for at least 6 months and will have viral loads less than 3,000 copies/ml. Participants in both cohorts will have blood drawn at study entry and Weeks 12 and 24. Blood samples will be used for CD4/CD8 cell count, plasma HIV-1 RNA, and immunologic assays.

ELIGIBILITY:
Inclusion Criteria for Cohorts A and B:

* HIV-1 infection
* CD4 cell count > 300 cells/mm3 within 60 days prior to study entry
* Negative pregnancy test within 14 days of starting study
* Agree to use acceptable methods of contraception while in study

Inclusion Criteria for Cohort A (Stable HAART) Only:

* Stable HAART regimen, defined as the suppression of viral load to undetectable levels, for at least 9 months prior to study entry
* Viral load < 75 copies/ml on at least three occasions within 9 months prior to study entry, with at least one of these values obtained between 6 and 9 months prior to study entry
* No single viral load >= 75 copies/ml within 9 months prior to study entry

Inclusion Criteria for Cohort B (Efficient Immune Control) Only:

* Not taking any antiretroviral drugs for at least 6 months prior to study entry
* Meets study definition of efficient immune control (generally HIV-1 viral load < 3,000 copies/ml, with some exceptions)

Exclusion Criteria:

* Pregnancy or breast-feeding
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements
* History of an AIDS-defining opportunistic infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54

CONTACTS AND LOCATIONS:
Overall Officials: R. Pat Bucy, MD, PhD, Study Chair — University of Alabama at Birmingham
Locations (6):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UC Davis Medical Center, Sacremento, California
  - University of Miami, Miami, Florida
  - Rush-Presbyterian/St. Lukes, Chicago, Illinois
  - Case Western Reserve University, Cleveland, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Bucy RP, Kilby JM. Perspectives on inducing efficient immune control of HIV-1 replication--a new goal for HIV therapeutics? AIDS. 2001 Feb;15 Suppl 2:S36-42. doi: 10.1097/00002030-200102002-00007. PMID 11424975
- [Background] Bucy RP. Immune clearance of HIV type 1 replication-active cells: a model of two patterns of steady state HIV infection. AIDS Res Hum Retroviruses. 1999 Feb 10;15(3):223-7. doi: 10.1089/088922299311394. No abstract available. PMID 10052752
- [Background] Pantaleo G, Menzo S, Vaccarezza M, Graziosi C, Cohen OJ, Demarest JF, Montefiori D, Orenstein JM, Fox C, Schrager LK, et al. Studies in subjects with long-term nonprogressive human immunodeficiency virus infection. N Engl J Med. 1995 Jan 26;332(4):209-16. doi: 10.1056/NEJM199501263320402. PMID 7808486
- [Result] Macatangay BJ, Zheng L, Rinaldo CR, Landay AL, Pollard RB, Pahwa S, Lederman MM, Bucy RP. Comparison of immunologic assays for detecting immune responses in HIV immunotherapeutic studies: AIDS Clinical Trials Group Trial A5181. Clin Vaccine Immunol. 2010 Sep;17(9):1452-9. doi: 10.1128/CVI.00498-09. Epub 2010 Jul 14. PMID 20631337